CLINICAL TRIAL: NCT01455649
Title: A Prospective, Open-label, Controlled, Randomized Study to Evaluate the Safety and Efficacy of Switching Calcineurin Inhibitor to Everolimus After 90 to 150 Days After Kidney Transplantation in Adults, Maintaining Corticosteroid and Mycophenolate Sodium Compared to Patients Who Will Maintain the Use of Calcineurin Inhibitor
Brief Title: Study to Evaluate the Safety and Efficacy of Switching Calcineurin Inhibitor to Everolimus After Kidney Transplantation in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Deise de Boni Monteiro de Carvalho (Other)
Responsible Party: Sponsor-Investigator, Deise de Boni Monteiro de Carvalho, Organ Transplant Technical Manager, Hospital Federal de Bonsucesso
Organization: Hospital Federal de Bonsucesso (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ABR17T
Record Dates: First submitted 2011-10-11; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Kidney Transplant; Immunosuppression
Keywords: Kidney; Transplant; Immunosuppression; Everolimus; Graft function
MeSH Terms: interventions — Everolimus; Calcineurin Inhibitors; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental)
  Interventions: Drug: Everolimus
- calcineurin inhibitor (Active Comparator)
  Interventions: Drug: calcineurin inhibitor

INTERVENTIONS:
Drug: Everolimus — Group will switch calcineurin inhibitor to everolimus within 1 day (overnight).
  Other Names: Certican
  Arms: Everolimus
Drug: calcineurin inhibitor — Group will maintain their initial immunosuppression therapy with calcineurin inhibitor
  Other Names: Tacrolimus, Cyclosporin, NeoOral, Prograf
  Arms: calcineurin inhibitor

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety in the use of everolimus, with its onset after 3 months of treatment with calcineurin inhibitor.

DETAILED DESCRIPTION:
The patient who met the inclusion and exclusion criteria will be included in the study and randomized into two groups in the third month post transplant, they will be in use of tacrolimus, corticosteroids and Mycophenolate sodium. The group 1 will undergo a conversion from calcineurin inhibitor to Everolimus within 1 day (overnight), group 2 will be maintained with the initial immunosuppression. We will start Everolimus at 1 mg 2x/day and three days after the beginning we will adjust the dose by the serum levels, which will be kept in 6 to 10ng/dL. The doses of corticosteroids and Mycophenolate sodium will be retained. There will be performed renal biopsies at randomization and after 12 months. The glomerular filtration rate will be calculated monthly using the MDRD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 65 years old
* First transplantation recipients
* PRA < 30%
* Living or cadaveric donor
* Stable renal function
* Patients not pregnant or breastfeeding , where pregnancy is defined as the woman status from conception to gestation conclusion, through a positive beta hCG test (>5mUI/mL)
* Provided written informed consent form

Exclusion Criteria:

* Cadaveric donor with expanded criterion
* Multiple organs transplantation
* Kidney cold ischemia time > 24 hours
* Severe rejection episode - Banf >IIA
* Glomerular filtration rate < 35mL/min
* Presence of hard to treat dyslipidemia - severe hypercholesterolemia (>350mg/dL) or hypertriglyceridemia (>500mg/dL)
* Proteinuria > 800mg/24h
* Patients with history of malignancy of any organic system, treated or not, within 5 years, with or without evidence of local recurrence or metastases, other than localized basal cell carcinoma
* Female with childbearing potential without using a reliable contraceptive method.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Creatinine Clearance at 24 months | baseline and two years
  The primary objective is to demonstrate the effectiveness and non-inferiority of treatment with everolimus, by assessing renal function, in comparison with the use of calcineurin inhibitor.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | baseline and two years
  The secondary objective is to demonstrate the safety by comparing rejection episodes, graft loss, infection, cancer and death in the control group

CONTACTS AND LOCATIONS:
Overall Officials: Francisco G Miloski, MD, Study Chair — Physician; Tereza Matuck, MD, Study Chair — Chief of the Nephrology Department; Regina Sousa, Study Chair — Head Nurse of The Nephrology Department
Locations (1):
- Hospital federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro, Brazil